CLINICAL TRIAL: NCT05380024
Title: A Study of Ensartinib as Neoadjuvant Therapy for Patients With ALK Positive Resectable Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wu Nan, Clinical Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-EN-IV0012
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Resectable; NSCLC; ALK-TKI; Ensartinb; Neoadjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ensaritinib (Experimental)
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — Ensartinib 225mg QD 8 weeks

SUMMARY:
This is a Phase II, single-Arm, prospective study of neoadjuvant Ensartinib for the treatment of patients with ALK positive, resectable for stage II to IIIB(N2) Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Male or female, at least 18 years of age.
* Histologically or cytologically documented lung adenocarcinoma within 60 days prior to study enrollment.
* Clinical stage IIA/IIB/IIIA/IIIB assessed by EBUS-TBNA or PET(positron emission tomography)/CT can be resected.
* Patients confirmed as ALK positive (FISH or Ventana IHC or RT-PCR, NGS)
* Presence of at least one accurately measurable lesion, CT showing a maximum diameter of 10mm at baseline (except for lymph nodes with a short axis of 15mm required) and suitable for accurate repeat measurements.
* Eastern Cooperative Oncology Group (ECOG) performance status （PS） of 0 or 1 at enrolment.
* Hematology , liver and kidney function are adequate for neoadjuvant therapy.
* Cardiopulmonary function suitable for surgical treatment (ECG, echocardiography, pulmonary function or blood gas analysis).
* Serum pregnancy test (for females of childbearing potential) negative at screening.Female patients of non-childbearing potential must meet at least 1 of the following criteria:

  ① Achieved postmenopausal status, defined as follows: cessation of regular menses forat least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle- stimulating hormone (FSH)level confirming the postmenopausal state;

  ② Have undergone a documented hysterectomy and/or bilateral oophorectomy;

  ③ Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations） are considered to be of childbearing potential.
* Male subjects must be willing to use barrier contraception

Exclusion Criteria:

* Mixed squamous cell carcinoma, large cell carcinoma，small cell lung cancer.
* Prior treatment with any systemic anti-cancer therapy for NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
* Pregnant female patients; breastfeeding female patients.
* Current use of (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of Cytochrome P450 3A4(CYP3A4)(at least 3 weeks prior).
* Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding, that the investigator considers to be detrimental to patient participation in the study or to adherence to the protocol. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C virus (HCV) (e.g., in case of known HBsAg or HCV antibody positivity), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
* Past medical history of Interstitial lung disease（ ILD）, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* A history of hypersensitivity to Icotinib with or without active excipients or to drugs of similar chemical structure or class, and uncontrollable nausea and vomiting, chronic gastrointestinal disease, inability to swallow formulated drugs, or having undergone major bowel resection that would interfere with adequate absorption of Ensartinib.
* Any of the following cardiac criteria:

  ①Mean resting corrected QT interval (QTc)>470 msec, obtained from 3 electrocardiograms (ECGs)

  ②Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250msec, symptomatic bradycardia <45 beats/minute.

  ③Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
* A clear past history of neurological or psychiatric disorders, including epilepsy or dementia;
* Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as ≤10% residual cancer cells in the main tumour, as assessed per central pathology laboratory post-surgery

SECONDARY OUTCOMES:
Pathological complete response (pCR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as absence of any residual cancer cells in the dissected tumour samples, including the main tumour and lymph nodes, assessed post-surgery
Objective response rate(ORR) | Baseline (Prior to surgery)
  ORR is defined as the percentage of participants having a complete response or a partial response, measured by RECIST 1.1.
Disease free survival (DFS) | From date of randomization up to approximately 42 months after date of resection
  DFS is defined as the time from the date of surgery until the first date of disease recurrence (local or distant) or date of death due to any cause, whichever occurs first.
Overall Survival (OS） | Up to approximately 5.5 years after the last patient is randomized
  Defined as the time from the date of entry to the date of death from any cause.
Incidence of Adverse Events | From the time of enrollment to either 28-days after the last dose of last study treatment for patients who do not undergo surgery, or 90-days post-surgery
  AE captured by CYCAE 5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - NAN Wu, Beijing, Beijing Municipality